CLINICAL TRIAL: NCT04741802
Title: Feasibility and Acceptability of a Community-based Weight Loss Program Among African American Breast Cancer Survivors
Brief Title: TOPS for African American Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00107615
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Feasibility and Acceptability of the TOPS Program; Obesity; Breast Cancer; Weight Loss
MeSH Terms: conditions — Obesity; Breast Neoplasms; Weight Loss | interventions — TOPS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOPS (Experimental): weight loss program (Take Off Pounds Sensibly, TOPS) for overweight and obese African American breast cancer survivors
  Interventions: Behavioral: TOPS

INTERVENTIONS:
Behavioral: TOPS — weight loss program (Take Off Pounds Sensibly, TOPS) for overweight and obese African American breast cancer survivors in the local chapter of a national African American breast cancer support group (Sisters Network Triangle North Carolina, SNTNC).

SUMMARY:
For women diagnosed with breast cancer, dietary, weight loss, and physical activity have been linked with clinically significant weight loss; decreased risk of death; reduced risk of breast cancer recurrence; fewer cardiovascular events; and improved physical function. The objectives of these aims are to a) determine if the TOPS materials and format are possible and accepted by overweight and obese African American breast cancer survivors; b) gather data for sample size calculations for a larger future study.

To meet these aims, we will collect data to see if participants enjoyed the TOPS program and suggestions for changes to the program to make it fit their needs. Other methods will measure recruitment, retention, and weight change.

Aim 1: Examine the feasibility and acceptability of a national, low-cost, community-based, peer-led, weight loss program (Take Off Pounds Sensibly, TOPS) for overweight and obese African American breast cancer survivors in the local chapter of a national African American breast cancer support group (Sisters Network Triangle North Carolina, SNTNC).

Aim 2: Assess the weight change of overweight and obese African American breast cancer survivors after 6 months in the TOPS program to gather data for sample size calculations for a future RCT (randomized controlled trial).

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer with BMI ≥ 25 kg/m after completion of primary 2 therapy (surgery, radiation, adjuvant or neo-adjuvant chemotherapy).

Exclusion Criteria:

* Women whose oncology providers do not agree with their participation in a weight loss program or those participating in another weight loss program.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nia Mitchell, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local chapter of a national African American breast cancer support group (Sisters Network Triangle North Carolina, SNTNC), which has a roster of 160 members.
Period: Overall Study
Arm/Group | TOPS
Started | 26
Completed | 14
Not Completed | 12
Not completed — Death | 1
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Arm/Group | TOPS
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Invited Women Who Attended the TOPS (Take Off Pounds Sensibly) Information Session
Time Frame: One-time invitation
Population: Women who were invited to attend the information session (all members of the Sisters Network Triangle North Carolina).
Measure: Count of Participants; unit: Participants
Arm/Group | TOPS
Number analyzed (Participants) | 160
Participants | 45

2. Primary Outcome: Number of Women Who Attended the Information Session and Joined the TOPS Program
Time Frame: One-time information session
Population: Number of women who attended the information session.
Measure: Count of Participants; unit: Participants
Arm/Group | TOPS
Number analyzed (Participants) | 45
Participants | 26

3. Primary Outcome: Number of Women Who Remained in the Program for 12 Weeks
Description: Measured by the number of women who reported to the 12-week weigh in.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TOPS
Number analyzed (Participants) | 26
Participants | 23

4. Primary Outcome: Number of Women Who Remained in the Program for 24 Weeks
Description: Measured by the number of women who reported to the 24-week weigh in.
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TOPS
Number analyzed (Participants) | 26
Participants | 18

5. Secondary Outcome: Percent Change in Participants' Weight as Measured by Scale Reading
Time Frame: baseline, 3 months, 6 months, 12 months
Population: Completers at each time point.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | TOPS
Number analyzed (Participants) | 23
percentage of change
  Baseline to 3 months | -2.6 (3.5)
  Baseline to 6 months: number analyzed (Participants) | 18
  Baseline to 6 months | -3.5 (4.5)
  Baseline to 12 months: number analyzed (Participants) | 14
  Baseline to 12 months | -6.4 (5.5)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | TOPS
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT04741802/Prot_001.pdf
  • Informed Consent Form (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT04741802/ICF_002.pdf